CLINICAL TRIAL: NCT04424563
Title: Activated Factor Seven (aFVII) Versus Aminocaproic Acid For Treatment of Traumatic Retro-Peritoneal Hematoma
Brief Title: Activated Factor Seven in Traumatic Retro Peritoneal Hematoma
Status: Completed | Type: Observational
Sponsor: King Abdul Aziz Specialist Hospital (Network)
Responsible Party: Sponsor
Other Study IDs: ICU-8-20
Record Dates: First submitted 2020-06-06; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2019-12

CONDITIONS: Traumatic Bleeding
MeSH Terms: interventions — Ventilators, Mechanical; Aminocaproic Acid; recombinant FVIIa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Group A: Patients of group A include 40 patients, received aminocaproic acid at dose of 4 gram slowly intravenous infusion over 1 hour and continues slowly intravenous infusion 1 gram/ hour for 8 hours.
  Interventions: Device: ventilators; Drug: aminocaproic acid
- Group B: While patients of group B include 40 patients, received aFVII according to the following protocol, First dose 200 microgram/kg. If patient still oozing, vital data not stable and/or could not achieve and keep the target Hb (>10 gm%) another 2 doses of aFVII received each dose 100microgram /kg 1 hour and 3 hours apart from the initial dose if needed.
  Interventions: Device: ventilators; Drug: Novo Seven

INTERVENTIONS:
Device: ventilators — all patients in both groups will be ventilated if shocked and no recordable blood pressure
Drug: aminocaproic acid — 4 gram slowly intravenous infusion over 1 hour and continues slowly intravenous infusion 1 gram/ hour for 8 hours.
  Other Names: Amicar
  Groups: Group A
Drug: Novo Seven — 200 microgram/kg. If patient still oozing, vital data not stable and/or could not achieve and keep the target Hb (>10 gm%) another 2 doses of aFVII received
  Other Names: activated factor seven
  Groups: Group B

SUMMARY:
80 patients with traumatic retro-peritoneal hematoma allocated into two groups 40 patients each. Patients of Group A received aminocaproic acid while patients of group B received aFVII. Number of packed RBCs given to get target Hb level and time to get this target Hb level (>10 gm%) recorded as indicators for control bleeding. Blood pressure, pulse, Arterial blood gasses and urine output recorded as indicator for treatment of hypovolemic shock. hypoxic index, chest X ray and coagulation profile used as indicator for complication.

DETAILED DESCRIPTION:
80 patients admitted to King Abdul-Aziz Specialist Hospital in Taif, KSA between May 2017 and December 2019 with polytrauma and severe retroperitoneal bleeding diagnosed by abdominal computerized tomography.

King Abdelaziz research and ethical committee approved the project under heading of ethical approval and heading of human and animal rights along with Helsinki Declaration.

A written consent from the patient or from their 1st degree relative was obtained if patient intubated. The primary outcome of This study divided into 3 parts. 1st 0ne compare the ability of both drugs to stop retroperitoneal bleeding efficiently and in shorter time for these 2 measurable indicators selected in our study the number of packed RBCS needed to achieve hemoglobin level (Hb) > 10 gm% and the time needed to achieve this target Hb. the 2nd part indicators divided into clinical indicators (blood pressure, pulse and urine output) and laboratory indicators [arterial blood gases especially PH, and bicarbonate concentration (HCO3)]. the 3rd part indicators PT, PTT and Platelets count were used as indicator for DIC and hypoxic index and chest x ray were used as indicator for TRALI (transfusion related acute lung injury).

Resuscitation done in all patients in both groups according to hospital protocol by crystalloid (normal saline), colloids [plasma protein fraction-packed RBCs, fresh frozen plasma], until achieve satisfactory stable vital data. All laboratory work samples were collected (CBC complete blood picture, Blood chemistry included liver enzymes and kidney function tests, Coagulation profile, arterial blood gasses).

Urine output collected hourly. Our study included any patient who received more than 50ml/kg blood during the first 8hours after admission in order to achieved a hemoglobin level >10 gram %, with platelet count more than 50, 000/mm3 after resuscitation and Their temperature was more than 36 degree centigrade after warming. Which considered criteria needed to get maximum effect from aFVII if used intravenously. Patient randomized into 2 groups, 40 patients in each, this done by randomization numbers. Patients of group A received aminocaproic acid at dose of 4 gram slowly intravenous infusion over 1 hour and continues slowly intravenous infusion 1 gram/ hour for 8 hours. While patients of group B received aFVII according to the following protocol, First dose 200 microgram/kg. If patient still oozing, vital data not stable and/or could not achieve and keep the target Hb (>10 gm%) another 2 doses of aFVII received each dose 100microgram /kg 1 hour and 3 hours apart from the initial dose if needed. The exclusion criteria in our study, if patient had cardiac arrest before giving aFVII, deeply comatose with Glasgow coma scale (GCS) 3/15 and pupil dilated fixed.

All patient in both groups observed for 48hours and the following indicators recorded.

Indicators for efficacy of stop bleeding (number of packed RBCs needed to keep hemoglobin level >10 gm% and time needed to reach this target Hb).

Indicators for ability of both drugs to treatment the hemorrhagic shock and restore tissue perfusion (and this assessed by clinical indicators blood pressure, pulse and urine output and laboratory indicators as arterial PH and bicarbonate concentration ( HCO3) Indicators for ability of both drugs to protect the patients with retroperitoneal hematoma from complications of massive blood transfusion and in this 2 complications were selected the disseminated intra-vascular coagulopathy (DIC) and PT, PTT, Platelets count were used as indicators and (TRALI) transfusion related acute lung injury and the hypoxic index and chest x ray were used as indicators. The duration of the study only two days and the data recorded every 8 hours.

ELIGIBILITY:
Inclusion Criteria:

* severe bleeding

Exclusion Criteria:

* post arrest

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 80 patients admitted to King Abdul-Aziz Specialist Hospital in Taif, KSA between May 2017 and December 2019 with polytrauma and severe retroperitoneal bleeding diagnosed by abdominal computerized tomography.
  King Abdelaziz research and ethical committee approved the project under heading of ethical approval and heading of human and animal rights along with Helsinki Declaration.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
stop bleeding | 2 days
  efficacy of activated factor seven with aminocaproic acid in medical treatment of retroperitoneal bleeding,

CONTACTS AND LOCATIONS:
Locations (1):
- King abd el Aziz specialist hospital, Ta'if, Saudi Arabia